CLINICAL TRIAL: NCT05606926
Title: Effect of Whole Body Vibration With Weighted Vest on Motor Function in Children With Spastic Diplegia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mahmoud Abd-elmonem, Assist Prof. Physiacl therapy for pediatric department, faculty of physical therapy , Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: whole body vibration
Record Dates: First submitted 2022-09-27; First posted 2022-11-07 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; balance; muscle strength; spastic diplegia; HUMAC balance system
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Other): 15 Children with spastic diplegia in this group will a designed physical therapy program for 60 minutes per session in addition to WBV for 10 minutes, three times a week, for three consecutive months.
  Interventions: Other: physical therapy program; Other: whole body vibration (without extra weight vest)
- Experimental group (Experimental): 15 Children with spastic diplegia in this group will receive the same designed physical therapy program while WBV will be conducted while wearing a weighted vest.
  Interventions: Other: physical therapy program; Other: whole body vibration (with weight vest)

INTERVENTIONS:
Other: physical therapy program — Flexibility exercises to restore joint mobility of soft tissues, Static and dynamic balance exercises, Functional gait training , Functional strengthening exercises will be conducted three times a week, for three consecutive months.
Other: whole body vibration (without extra weight vest) — 9 minutes of three sets of 3-min semi-squats on the vibration platform. three times a week, for three consecutive months.
  Arms: Group I
Other: whole body vibration (with weight vest) — The extra-weight applied in the vest will be calculated as 10% of the child body weight. The vest is designed to allow small bags of sand with different weights that are distributed equally on anterior-posterior and mediolateral plans.
  Arms: Experimental group

SUMMARY:
Whole body vibration has been widely used in rehabilitation of individuals with disabilities as well as children with cerebral palsy. Previous studies have demonstrated the efficacy of Whole body vibration on balance, gross motor function, spasticity and bone density in children with cerebral palsy. However, adding extra weight during Whole body vibration for children with cerebral palsy as a means of enhancing the potential effects of Whole body vibration is unknown. Therefore, the aim of this study is to examine the effect of Whole body vibration with weighted vest on trunk control, balance and gross motor function in children with spastic diplegia.

ELIGIBILITY:
Inclusion Criteria:

* Their age will range from 8-12 years, from both sexes.
* Level II and III of gross motor functional classification system
* Grade 1 and 1+ spasticity according to the Modified Ashworth Scale
* Ability to understand and follow simple verbal instruc

Exclusion Criteria:

* Uncontrolled epilepsy.
* Mental retardation or autistic features.
* Medication changes that could affect muscle strength or tone
* Significant visual or auditory problems according to medical reports (audio-vestibular and ophthalmic examination),
* Structural or fixed soft tissue deformities of the lower and/or upper extremities.
* Neurological or orthopedic surgery in the past 12 months in the lower and/or upper extremities.
* Botox injection in the lower and/or upper extremities in the past 6 months.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Trunk control | three months
  The Trunk Control Measurement Scale is used to assess trunk control and consists of static and dynamic sitting balance in children aged 8 to 15 years with spastic CP
Gross motor function | three months
  The Gross motor function measure-88 will be used to assess motor function in 88 items across five dimensions: (a) lying and rolling, (b) sitting, (c) crawling and kneeling, (d) standing, and (e) walking, running and jumping. dimensions D and E will be assessed in the current study The assessment of each item will be conducted carefully and scored according to the scale scoring key (scale from 0-3) with total score 100 and higher score represent better performance
balance | three months
  Human computer balance system will be used to assess balance to assess center op pressure and limits of stability

CONTACTS AND LOCATIONS:
Overall Officials: HOSAM A ALMOHANDES, B.S.C, Study Director — Cairo university, faculty of physical therapy; Nahla M Ibrahim, Phd, Study Chair — Cairo university, faculty of physical therapy